CLINICAL TRIAL: NCT04808037
Title: A Phase 1/2 Study of Belantamab Mafodotin in Combination With Lenalidomide and Dexamethasone in Transplant-ineligible Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Blmf, Lenalidomide and Dexamethasone in Transplant-ineligible Patients With Newly Diagnosed Multiple Myeloma
Acronym: BelaRd
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hellenic Society of Hematology (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAE-2020/MM0107
Record Dates: First submitted 2021-03-04; First posted 2021-03-19 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1, First Part (Experimental): 12 patients are anticipated to receive Belantamab Mafodotin 2.5 Q8W = 2.5 mg/kg on Day 1 of every other 28-day cycle, in combination with Lenalidomide and Dexamethasone
  Interventions: Drug: Belantamab mafodotin
- Cohort 2, First Part (Experimental): 12 patients are anticipated to receive Belantamab Mafodotin 1.9 Q8W = 1.9 mg/kg on Day 1 of every other 28-day cycle, in combination with Lenalidomide and Dexamethasone
  Interventions: Drug: Belantamab mafodotin
- Cohort 3, First Part (Experimental): 12 patients are anticipated to receive Belantamab Mafodotin 1.4 Q8W = 1.4 mg/kg on Day 1 of every other 28-day cycle, in combination with Lenalidomide and Dexamethasone
  Interventions: Drug: Belantamab mafodotin
- Group A, Second Part (Experimental): 15 patients are anticipated to receive Belantamab Mafodotin in the Recommended Phase 2 Dose, in combination with Lenalidomide and Dexamethasone.
  In this Arm the ocular toxicity will be graded according to the Dose Modification Guidelines for Corneal-Related Adverse Events Associated with belantamab mafodotin
  Interventions: Drug: Belantamab mafodotin
- Group B, Second Part (Experimental): 15 patients are anticipated to receive Belantamab Mafodotin in the Recommended Phase 2 Dose, in combination with Lenalidomide and Dexamethasone.
  In this Arm the ocular toxicity will be graded according to the Dose modification guidance based on visual acuity
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin in combination with Lenalidomide and Dexamethasone in patients with newly diagnosed Multiple Myeloma transplant-ineligible
  Other Names: Blenrep

SUMMARY:
This is a phase 1/2, open label, study designed to assess the safety and clinical activity of different Belantamab Mafodotin doses in combination with lenalidomide and dexamethasone.

DETAILED DESCRIPTION:
This is a phase 1/2, open label, study designed to assess the safety and clinical activity of different Belantamab Mafodotin doses in combination with lenalidomide and dexamethasone.

The study is comprised of two distinct parts: Part 1 will evaluate different doses of belantamab mafodotin in combination with lenalidomide and dexamethasone in up to 3 cohorts and will determine the recommended Phase 2 dose (RP2D) to be further evaluated for safety and clinical activity in the dose expansion cohort (Part 2). The RP2D dose will be used for future studies in the transplant-ineligible newly diagnosed MM setting. Part 2 of the study will also evaluate an alternative dose modification guideline for corneal adverse events.

Participants will undergo visits and assessments in accordance with the Schedule of Assessments (SoA).

Overall, approximately 66 participants will be enrolled in the study. Participant follow up will continue until 5 years after the last participant is randomized. The estimated accrual period will be 12 months corresponding to an approximate total study duration of 6 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participant at least 18 years of age
2. Monoclonal plasma cells in the bone marrow ≥10% or presence of a biopsy proven plasmacytoma and documented multiple myeloma satisfying at least one of the calcium, renal, anemia, bone (CRAB) criteria or biomarkers of malignancy criteria:

   CRAB criteria:

   i. Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than upper limit of normal (ULN) or >2.75 mmol/L (>11 mg/dL).

   ii. Renal insufficiency: creatinine clearance <40mL/min or serum creatinine >177 μmol/L (>2 mg/dL).

   iii. Anemia: hemoglobin >2 g/dL below the lower limit of normal or hemoglobin <10 g/dL.

   iv. Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET-CT.

   Biomarkers of Malignancy:
   1. Clonal bone marrow plasma cell percentage ≥60%.
   2. Involved: uninvolved serum FLC ratio ≥100.
   3. >1 focal lesion on magnetic resonance imaging (MRI) studies.
3. Must have at least ONE aspect of measurable disease, defined as one of the following:

   * Urine M-protein excretion ≥200 mg/24 hrs (≥0.2g/24 hrs), or
   * Serum M-protein concentration ≥0.5 g/dL (≥5.0 g/L), or
   * Serum free light chain (FLC) assay: involved FLC level ≥10 mg/dL (≥100 mg/L) and an abnormal serum free light chain ratio (<0.26 or >1.65).
4. Not a candidate for high-dose chemotherapy with ASCT due to presence of significant comorbid condition(s), such as cardiac, pulmonary or other major organ dysfunction that are likely to have a negative impact on tolerability of high dose chemotherapy with stem cell transplantation, as judged by the investigator. The reason(s) for transplant ineligibility will be collected in the case report forms (CRFs).
5. ECOG status of 0-2 (see Appendix 1).
6. Adequate organ system function as defined by the below laboratory assessments. Hematologic

   * Absolute neutrophil count (ANC) ≥1.5 X 109/L; GCSF use is NOT allowed to reach this level.
   * Hemoglobin ≥ 8.0 g/dL; transfusions are permitted.
   * Platelet count ≥ 50 x 109/L if bone marrow is >50% involved in myeloma. Otherwise ≥75 x 109/L; transfusions are NOT allowed to reach this level.

   Hepatic
   * Total bilirubin ≤1.5X ULN (Isolated bilirubin ≥1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
   * ALT ≤ 2.5 X ULN. Renal
   * eGFR ≥30 mL/min/1.73 m2; calculated using the Modified Diet in Renal Disease (MDRD) formula.
   * Spot urine (albumin/creatinine ratio) <500 mg/g (56 mg/mmol) OR
   * Urine Dipstick: Negative trace; if ≥1+ only eligible if confirmed <500 mg/g [56 mg/mmol] by albumin/creatinine ratio (spot urine from first void).
7. Female participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies:

   A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
   * Is not a woman of childbearing potential (WOCBP) OR
   * Is a WOCBP and using two methods of reliable birth control (one method that is highly effective and one additional effective [barrier] method), beginning 4 weeks prior to initiating treatment with lenalidomide, during therapy, during dose interruptions and continuing for 4 weeks following discontinuation of lenalidomide treatment. Thereafter, WOCBP participants must use one method of reliable birth control that is highly effective for a further 3 months following discontinuation of belantamab mafodotin. WOCBP must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction during treatment, during dose interruptions and for 28-days following the last dose of lenalidomide or 4 months following discontinuation of belantamab mafodotin treatment whichever is longer. For contraception guidance please refer to Appendix 2.

   A WOCBP must have two negative pregnancy tests prior to initiating therapy. The first test should be performed within 10-14 days and the second test within 24 hours prior to the start of lenalidomide therapy.

   The participant should not receive lenalidomide until the investigator has verified that the results of these pregnancy tests are negative. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.

   WOCBP is a female who:
   * has achieved menarche at some time point
   * has not undergone a hysterectomy or bilateral oophorectomy or
   * has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
8. Male participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies:

   Male participants are eligible to participate if they agree to the following during the intervention period and until 28 days after the last dose of lenalidomide or 6 months after the last dose of belantamab mafodotin, whichever is longer, to allow for clearance of any altered sperm.

   • Refrain from donating sperm

   PLUS either:
   * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, OR
   * Must agree to use contraception/barrier as detailed below:

   Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females).
9. Participants must be able to understand the study procedures and agree to participate in the study by providing written informed consent.

Exclusion Criteria:

-

Participants are excluded from the study if any of the following criteria apply:

1. Prior systemic therapy for multiple myeloma, or SMM.

   * NOTE 1: An emergency course of steroids (defined as no greater than 40 mg of dexamethasone, or equivalent per day for a maximum of 4 days (that is, a total of 160 mg) is permitted.
   * NOTE 2: Focal palliative radiation is permitted prior to enrollment, provided that it occurred at least 2 weeks prior to the first dose of study drug, that the participant has recovered from radiation-related toxicities, and that the participant did not require corticosteroid administration (for a longer period than that specified in NOTE 1 above) for radiation-induced adverse events
2. Participant is eligible for high dose chemotherapy with ASCT, as determined by a frailty score of 0 as assessed by the IMWG frailty index (1).
3. Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the NCI CTCAE Version 5.
4. Major surgery within 4 weeks prior to the first dose of study drug.
5. Presence of active renal condition (infection, requirement for dialysis or any other significant condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfil the other inclusion criteria.
6. Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
7. Evidence of active mucosal or internal bleeding uncontrolled by local therapy and not explained by reversible coagulopathy.
8. Current active liver or biliary disease (except for Gilbert's syndrome or asymptomatic gallstones, or otherwise stable chronic liver disease as per the Investigator's assessment).
9. Participants with previous or concurrent malignancies other than multiple myeloma are excluded. Exceptions are surgically treated cervical carcinoma in situ, or any other malignancy that has been considered medically stable for at least 2 years. The participant must not be receiving active therapy, other than hormonal therapy for this disease.

   o Note: Participants with curatively treated non-melanoma skin cancer are allowed without a 2-year restriction.
10. Evidence of cardiovascular risk including any of the following:

    * Evidence of current clinically significant untreated arrhythmias, including clinically significant ECG abnormalities, second degree (Mobitz Type II) or third degree atrioventricular (AV) block.
    * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of Screening.
11. Class III or IV heart failure as defined by the New York Heart Association functional classification system (Appendix 3).
12. Uncontrolled hypertension.
13. Active infection requiring treatment.
14. Known HIV infection, unless the participant can meet all of the following criteria:

    * Established anti-retroviral therapy (ART) for at least 4 weeks and HIV viral load <400 copies/mL.
    * CD4+ T-cell (CD4+) counts ≥350 cells/uL.
    * No history of AIDS-defining opportunistic infections within the last 12 months. o Note: consideration must be given to ART and prophylactic antimicrobials that may have a drug:drug interaction and/or overlapping toxicities with belantamab mafodotin or other combination products as relevant (See Section 7.2, Drug Interactions)
15. To be seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]).

    * Note 1: Participants with resolved infection (i.e., participants who are positive for antibodies to hepatitis B core antigen [antiHBc] or antibodies to hepatitis B surface antigen [antiHBs]) must be screened using real-time polymerase chain reaction (PCR). Those who are PCR positive will be excluded.
    * Note 2: presence of antiHBs indicating previous vaccination will not constitute an exclusion criterion.
16. Positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment unless the participant can meet the following criteria:

    * RNA test negative
    * Successful anti-viral treatment (usually 8 weeks duration) is required, followed by a negative HCV RNA test after a washout period of at least 4 weeks.
17. Current corneal epithelial disease except for mild punctate keratopathy.

    o Note: Participants with mild punctate keratopathy are allowed.
18. Intolerance or contraindications to anti-viral prophylaxis.
19. Unable to tolerate antithrombotic prophylaxis.
20. AL amyloidosis (light chain amyloidosis), active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma proliferative disorder, skin changes) or active plasma cell leukemia at the time of screening.
21. Exhibiting clinical signs of or has a known history of meningeal or central nervous system involvement by multiple myeloma.
22. Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
23. Use of an investigational drug within 14 days or five half-lives (whichever is longer) preceding the first dose of study drug.
24. Plasmapheresis within 7 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2028-09-08 (Estimated); Study Completion 2028-11-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) in each of the cohorts 1-3 | Five (5) years after last participant randomization
  Determination of the safety and tolerability of belantamab mafodotin in combination with lenalidomide and dexamethasone to establish a recommended Phase 2 dose for participants with newly diagnosed Multiple Myeloma, transplant-ineligible
Overall Response rate as per IMWG by Investigator Assessment, defined as the percentage of participants with a confirmed PR, VGPR, CR or sCR | Five (5) years after last participant randomization
  Evaluation of the preliminary clinical activity of the Recommended Phase 2 Dose of belantamab mafodotin in combination with lenalidomide and dexamethasone for participants with newly diagnosed Multiple Myeloma, transplant-ineligible
Number of participants with adverse events (AEs) and serious adverse events (SAEs) in each of the cohorts 1-3 | Five (5) years after last participant randomization
  Determine the safety and tolerability of blmf in combination with lenalidomide and dexamethasone to establish a recommended Phase 2 dose for participants with newly diagnosed Multiple Myeloma, transplant-ineligible
Number of participants with adverse events (AEs) and serious adverse events (SAEs) in patients receiving the Recommended Phase 2 Dose | Five (5) years after last participant randomization
  Further evaluation of the safety of Belantamab Mafodotin in combination with Lenalidomide and Dexamethasone

CONTACTS AND LOCATIONS:
Overall Officials: Meletios-Athanasios Dimopoulos, Principal Investigator — National and Kapodistrian University of Athens School of Medicine, Athens - Greece
Locations (1):
- General Hospital of Athens "Alexandra", Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gavriatopoulou M, Ntanasis-Stathopoulos I, Malandrakis P, Fotiou D, Migkou M, Theodorakakou F, Spiliopoulou V, Kanellias N, Eleutherakis-Papaiakovou E, Roussou M, Psarros G, Kastritis E, Dimopoulos MA, Terpos E. Belantamab mafodotin, lenalidomide, and dexamethasone in transplant-ineligible patients with newly diagnosed multiple myeloma: Analysis of belantamab mafodotin-associated ocular adverse events and their impact on daily functioning from the part 1 of a phase 1/2 study. Am J Hematol. 2024 Mar;99(3):502-504. doi: 10.1002/ajh.27219. Epub 2024 Jan 25. No abstract available. PMID 38270219